CLINICAL TRIAL: NCT06008535
Title: 10-year Results of Open Inguinal Hernia Repair. A Prospective Study
Brief Title: 10-year Results of Open Inguinal Hernia Repair
Status: Completed | Type: Observational
Sponsor: Tartu University Hospital (Other)
Responsible Party: Principal Investigator, Ceith Nikkolo, general surgeon, Tartu University Hospital
Other Study IDs: TartuUH_Surgery Clinic
Record Dates: First submitted 2023-07-18; First posted 2023-08-23 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Recurrence; Chronic Pain
MeSH Terms: conditions — Recurrence; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Open inguinal hernia repair — Lichtenstein hernioplasty or open inguinal hernia repair with self-gripping mesh

SUMMARY:
The main goal of the research is to evaluate the long-term results of open anterior alloplasty of inguinal hernia, mainly the occurrence of recurrences. The secondary aim of the study is to clarify the incidence of chronic pain and foreign body sensation 10 years after inguinal hernia surgery.

Patients who meet the criteria for inclusion in the study are invited to an appointment, where a questionnaire is filled out, an clinical examination and an ultrasound examination are performed.

ELIGIBILITY:
Inclusion Criteria:

* primary inguinal hernia operated between 2008-2013 at the Tartu University Hospital
* elective surgery
* age at least 18 years old at the time of the operation
* ability to understand the guidelines and willing to participate in the study

Exclusion Criteria:

* recurrent hernia
* strangulated hernia
* age under 18 years at the time of surgery
* does not agree to participate in the study
* does not understand the guidelines. Regarding the last exclusion criterion: since it is an assessment of the remote results of the treatment and probably relatively many of the subjects are very elderly, it may happen that when contacting the patient by phone it turns out that the patient is no longer adequate to make a decision about participating in the study or to answer questions (experienced cerebral infarction, dementia, etc. .) - in this case, the patient is not invited to the appointment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group consists of patients who were operated on with a primary inguinal hernia in the department of general surgery and plastic surgery between 2008-2013 at the Tartu University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Recurrence | at 10-year follow-up
  Inguinal hernia recurrence on clinical examination or in ultrasound

SECONDARY OUTCOMES:
Chronic pain | at 10-year follow-up
  Chronic pain after open inguinal hernia repair. The pain questionnaire includes questions about pain at rest, on coughing, when rising from lying to sitting position and during physical effort and exercise (yes-or-no questions). If the answer to these questions are positive, then the pain is measured on visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ceith Nikkolo, PhD, Principal Investigator — Tartu University Hospital
Locations (1):
- Tartu University Hospital, Tartu, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nikkolo C, Lillsaar T, Vaasna T, Kirsimagi U, Lepner U. Ten-Year Results of Inguinal Hernia Open Mesh Repair. J Abdom Wall Surg. 2025 Jun 9;4:14384. doi: 10.3389/jaws.2025.14384. eCollection 2025. PMID 40551961